CLINICAL TRIAL: NCT01763177
Title: Use of Oxygen Nebulizer for Preventing Post-operative Sore Throat
Acronym: POST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Panthila Rujirojindakul, Assistant Professor Dr.Panthila Rujirojindakul, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EC56-008-08-1-1
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Pain, Postoperative
Keywords: nebulizer; oxygen; post-operative sore throat
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No oxygen (No Intervention): No given oxygen at post-anesthetic care unit
- Oxygen (Active Comparator): Oxygen nebulizer via face mask, Fraction of inspired oxygen (FiO2) 0.4, flow 8 liter per minute (LPM) for 30 minutes
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Oxygen — Oxygen mask 40% 8 LPM for 30 minutes
  Arms: Oxygen

SUMMARY:
Rationale: Delivery dry gas during anesthesia is associated with post-operative sore throat (POST). Oxygen nebulizer therapy increases humidity to the airway, especially post-extubation.

Objective: To investigate the effect and complications of oxygen nebulizer therapy on POST.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Pre-operative Hb >10 g% or Hct > 30%
* American Society of Anesthesiologist (ASA) class I-III
* Elective surgery
* General anesthesia with oroendotracheal tube using Macintosh laryngoscope
* Not exposed to intraoperative nitrous oxide
* Oxygen saturation at room air > 95% before induction and at arrival the PACU

Exclusion Criteria:

* Cases needing ICU admission immediately post-operative
* Conditioning requiring post-operative oxygen therapy e.g. heart disease, pregnancy, morbid obesity, cardiac and thoracic surgery
* Patients' conditioning affecting to complication of nebulizer oxygen therapy e.g. pulmonary disease, bleomycin treatment
* Patient's conditioning affecting POST assessment e.g. pre-operative using ventilator, recent upper respiratory tract infection (URI), recent lower respiratory tract infection and history of difficult airway
* Surgical conditioning affecting POST e.g. airway surgery, oral surgery, esophageal and neck surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The effect of oxygen nebulizer therapy on post-operative sore throat | at post-anesthetic care unit and 24-h post-operative
  Assess POST using scoring system and discomfort by interview. Sore throat scoring system is divided into 4 scores 0 means no sore throat
  1. means minimal sore throat (less severe than cold)
  2. means moderate sore throat (similar to cold)
  3. means severe sore throat (more severe than cold)

SECONDARY OUTCOMES:
To evaluate the adverse events (pulmonary complications, wound infection, and mortality) of post-operative complications related to oxygen therapy | 24-h post-op and 30-d mortality

CONTACTS AND LOCATIONS:
Overall Officials: Panthila Rujirojindakul, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Prince of Songkla University
Locations (1):
- Department of anesthesiology, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Background] oxygen nebulizer AND sore throat
- See also: oxygen nebulizer AND sore throat — http://www.ncbi.nlm.nih.gov/pubmed/